CLINICAL TRIAL: NCT06860776
Title: Pilot Study on the Analysis of the Metabolic Phenotype in Individuals With Difficulties in Losing and Gaining Weight
Brief Title: How Metabolism Affects Weight Loss and Gain
Status: Recruiting | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Tim Hollstein, Principal Investigator, University Hospital Schleswig-Holstein
Other Study IDs: D 481/24
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Obesity and Overweight
Keywords: obesity; metabolic phenotype; thrifty; spendthrift; diet-induced thermogenesis; fasting; indirect calorimetry
MeSH Terms: conditions — Obesity; Overweight; Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Urine, Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lean individual with weight gain difficulties: Participants in this group are lean individuals (BMI 18.5-22.0 kg/m²) who have difficulty gaining weight. They will undergo a 24-hour fasting period followed by a controlled low-protein, high-calorie meal test. Researchers will measure their resting metabolic rate before and after fasting, as well as the body's response to the test meal. By comparing these results to those of other groups, the study aims to identify metabolic factors that influence weight gain difficulties and guide future personalized treatments.
- Individuals with obesity and weight loss difficulties: Participants in this group are individuals with obesity (BMI >30 kg/m²) who have difficulty losing weight. They will undergo a 24-hour fasting period followed by a controlled low-protein, high-calorie meal test. Researchers will measure their resting metabolic rate before and after fasting, as well as the body's response to the test meal. By comparing these findings with those of other groups, the study seeks to uncover metabolic factors that contribute to weight loss difficulties and guide more personalized treatment approaches.

SUMMARY:
This study examines why some individuals with obesity have difficulty losing weight, whereas some lean individuals struggle to gain weight. The investigators will measure how the human body uses energy during a fasting period and after consumption of a specially designed, low-protein meal. By comparing these responses, the investigators aim to identify different "metabolic phenotypes" that affect weight control. Findings from this research may lead to more personalized treatments for managing weight. Participation in this study involves simple tests and basic body measurements.

DETAILED DESCRIPTION:
This study aims to better understand why certain individuals find it difficult to lose weight while others struggle to gain weight. Investigators believe that differences in how the human body uses energy-referred to as the metabolic phenotype-may play a key role.

Two groups of participants will be compared: one group includes lean individuals who have difficulty gaining weight, and the other group consists of individuals with obesity who have difficulty losing weight. Participants will undergo a series of tests designed to measure how the human body burns calories under different conditions.

The study involves two main components:

1. 24-Hour Fasting Period: Participants will abstain from eating for 24 hours to observe how the body adapts by either conserving or maintaining energy expenditure.
2. Meal Test: Following the fasting period, participants will consume a specially designed, low-protein meal that simulates overeating. The investigators will measure how much additional energy is burned during digestion, a process known as diet-induced thermogenesis.

A technique called indirect calorimetry will record oxygen consumption and carbon dioxide production. These measurements help calculate resting energy expenditure (REE), which refers to the calories the body burns while at rest, and any changes that occur after fasting and eating.

The goal is to identify distinct metabolic patterns. Some individuals may have a "thrifty" metabolism that conserves energy, making weight loss more challenging, whereas others may have a "spendthrift" metabolism that expends more energy, potentially explaining difficulty in gaining weight. Understanding these differences could lead to more personalized and effective weight management strategies.

This study is conducted under strict safety and ethical standards to ensure minimal risk to participants. By examining the relationship between metabolism and weight control, the findings may pave the way for improved treatments for obesity and related weight issues.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 (Lean): BMI 18.5-22.0 kg/m², reporting difficulty gaining weight
* Group 2 (Obese): BMI >30 kg/m², reporting difficulty losing weight
* Healthy status as determined by medical history, physical examination, and laboratory tests
* Stable weight (less than 5% fluctuation) over the past 6 months

Exclusion Criteria:

* Prediabetes (HbA1c >5.6% or fasting blood glucose >100 mg/dL) or diabetes mellitus
* Conditions affecting appetite or energy expenditure (e.g., Cushing's syndrome, uncontrolled hyper-/hypothyroidism)
* Gastrointestinal disorders that impact nutrient absorption (e.g., inflammatory bowel disease, malabsorption syndromes, ulcers)
* Psychiatric conditions influencing eating behavior (e.g., active depression, anorexia nervosa, bulimia nervosa, borderline personality disorder)
* Acute, unstable cardiovascular disease requiring hospitalization within the last 6 months (e.g., stent placement)
* Cancer that required treatment in the past 5 years
* Chronic kidney disease (Stage IV or higher, per NKF criteria)
* Active infectious disease (e.g., HIV, hepatitis)
* Current nicotine use or nicotine use within the last month prior to screening
* Illicit drug use (e.g., amphetamines, cocaine, heroin, marijuana)
* Regular high-intensity physical activity (≥1 hour/day)
* Non-MRI-compatible metallic implants (e.g., artificial joints, metal plates)
* Pregnancy or breastfeeding
* Use of weight-loss medications
* Clinically significant claustrophobia
* Any other condition not mentioned above that, in the opinion of the investigator, could interfere with study participation or compromise patient safety

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the general adult population, focusing on two specific groups:
  1. Lean individuals (BMI 18.5-22.0 kg/m²) who struggle to gain weight
  2. Individuals with obesity (BMI >30 kg/m²) who struggle to lose weight
  All participants must be generally healthy, between 18 and 70 years old, and report a stable body weight (less than 5% fluctuation) in the last six months. Recruitment will occur via community outreach, advertisements, and existing volunteer registries. Potential participants with conditions or circumstances that could affect appetite, energy expenditure, or study compliance will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Identification of Metabolic Phenotypes in Lean vs. Obese Individuals | Measured at baseline (Day 1) and after 24-hour fasting (Day 2)
  We aim to determine whether individuals with obesity (BMI >30 kg/m²) exhibit a more "thrifty" metabolic phenotype (lower resting metabolic rate [RMR] after 24-hour fasting and reduced diet-induced thermogenesis [DIT]) compared to lean individuals (BMI 18.5-22 kg/m²) who have trouble gaining weight, hypothesized to show a more "spendthrift" metabolic phenotype (increased RMR after fasting and higher DIT). RMR is measured via indirect calorimetry before and after a 24-hour fast, followed by a high-calorie, low-protein meal test to assess DIT.

SECONDARY OUTCOMES:
Correlation Between Fasting-Induced Energy Expenditure Changes and Diet-Induced Thermogenesis | Baseline (Day 1), post-fasting (Day 2), and after the meal test (Day 2)
  Evaluate how the change in resting metabolic rate (RMR) after a 24-hour fast relates to diet-induced thermogenesis (DIT) following a high-calorie, low-protein meal. This will clarify the interaction between fasting adaptation and meal-related energy expenditure in lean vs. obese individuals.
Assessment of Metabolic Flexibility via Respiratory Quotient | Baseline (Day 1), post-fasting (Day 2), and after the meal test (Day 2)
  Determine whether individuals with obesity show a smaller shift in their respiratory quotient (RQ) after fasting and the meal test, indicating lower metabolic flexibility compared to lean participants.
Correlation Between Weight Gain at 12-Month Follow-Up and Initial Metabolic Phenotype | 12-month follow-up
  Body weight (in kilograms) will be measured at baseline and again after 12 months using a calibrated scale. The correlation between weight change over this period and the initial metabolic phenotype (classified as "thrifty" or "spendthrift") will be assessed. The metabolic phenotype is determined by changes in resting metabolic rate (RMR) and diet-induced thermogenesis (DIT), both measured via indirect calorimetry.
Correlation Between Weight Gain at 12-Month Follow-Up and Diet-Induced Thermogenesis | 12-month follow-up
  Body weight (in kilograms) will be measured at baseline and again after 12 months using a calibrated scale. The correlation between weight change over this period and the magnitude of diet-induced thermogenesis (DIT) will be assessed. DIT is determined via indirect calorimetry after a controlled, low-protein meal. This assessment will help identify whether higher or lower DIT predicts long-term weight change.
Correlation Between Meal Test Diet-Induced Thermogenesis and Fibroblast Growth Factor 21 (FGF-21) Secretion | After the meal test (Day 2)
  Fibroblast Growth Factor 21 (FGF-21) levels (in picograms per milliliter) will be measured in blood samples collected after the high-calorie, low-protein meal. The correlation between FGF-21 levels and diet-induced thermogenesis (DIT) will be assessed. DIT is measured using indirect calorimetry to quantify energy expenditure following the meal. This analysis will help determine whether FGF-21 may serve as a biomarker of metabolic adaptation.
Correlation Between Gut Hormones and Changes in Energy Expenditure | Baseline (Day 1), after 24-hour fast (Day 2), and after the meal test (Day 2)
  Serum levels of gut hormones (e.g., ghrelin, glucagon-like peptide-1 [GLP-1]) will be measured in picograms per milliliter. Resting metabolic rate (RMR) and diet-induced thermogenesis (DIT) will be assessed via indirect calorimetry before and after a 24-hour fast, as well as after a high-calorie, low-protein meal. The correlation between gut hormone levels and changes in energy expenditure (RMR and DIT) will be evaluated to investigate hormonal influences on metabolic responses.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Schleswig-Holstein, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study Website (German) — https://www.uksh.de/diabetologie-kiel/Forschung/Kohortenstudien/Pilotstudie+Stoffwechseltyp.html